CLINICAL TRIAL: NCT06842719
Title: Effectiveness of Post-Hospital Discharge Housing Counselling to Support Geriatric Patients in Staying At Home: a Pragmatic Randomised Controlled Trial
Acronym: Frail@Home
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maximilian König (Other)
Responsible Party: Sponsor-Investigator, Maximilian König, Prof. Dr., University Medicine Greifswald
Organization: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BB 079/24
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Frailty Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (on-site housing counseling) (Experimental): standard care plus an additional information booklet
  Interventions: Procedure: on-site housing counseling
- Control group (standard care plus an additional information booklet ) (No Intervention): standard care plus an additional information booklet

INTERVENTIONS:
Procedure: on-site housing counseling — on-site housing counseling by a certified housing counseling expert
  Arms: Intervention (on-site housing counseling)

SUMMARY:
Hospitalisation is often a disruptive event for older people, especially for geriatric patients with frailty. A critical factor for a successful return to one's own home is the living situation. Unfortunately, a large proportion of homes in Germany are not sufficiently accessible and often do no longer meet the needs of older residents with various health limitations. This can impair residents' functionality, increase the risk of falls, and restrict independence. Through timely housing advice and adaptation, including digital aids, more older people could be enabled to remain in their own homes with a high degree of safety despite their limitations ("Aging in Place").

Whilst long-term care insurance provide funding for home environment improvements, this is often not utilised, in part due to a lack of advice. The effectiveness of housing counselling in stabilising the functional level of geriatric patients after hospital discharge and in preventing negative outcomes such as rehospitalisation, falls, nursing home placement or death has not been sufficiently investigated in the German health and social care system. The few available studies show that interventions related to the home environment can have positive effects on activities of daily living, fall risk and mental health. As the functional abilities of older patients are usually worse at the time of discharge than before hospitalisation, this is a good time to assess the home environment and the person-environment fit.

Integrating professional housing counselling into discharge management could make a significant contribution to increasing safety in the home environment, improving self-help skills and preventing falls and re-hospitalisation. This could improve quality of life and reduce the burden on the healthcare system. The Frail@Home trial is a single-centre, randomised, controlled pragmatic trial (RCT) to test whether housing counselling provided within two to four weeks of hospital discharge increases the chances of older people remaining in their familiar home environment. The intervention group will receive on-site housing counseling, while the control group will receive standard care plus an additional information booklet from the local housing counseling service. The primary endpoint of the study is the number of days spent at home (DSH) in the first 6 and 12 months after discharge from acute geriatric care. The follow-up period will be 12 months. If successful, this study will be the first to show, using RCT methods, that early housing counselling after hospital discharge supports the retention of geriatric patients in their familiar homes.

DETAILED DESCRIPTION:
Hospitalisation is often a disruptive event for older people, especially for geriatric patients with frailty. A critical factor for a successful return to one's own home is the living situation. Unfortunately, a large proportion of homes in Germany are not sufficiently accessible and often do no longer meet the needs of older residents with various health limitations. This can impair residents' functionality, increase the risk of falls, and restrict independence. Through timely housing advice and adaptation, including digital aids, more older people could be enabled to remain in their own homes with a high degree of safety despite their limitations ("Aging in Place").

Whilst long-term care insurance provide funding for home environment improvements, this is often not utilised, in part due to a lack of advice. The effectiveness of housing counselling in stabilising the functional level of geriatric patients after hospital discharge and in preventing negative outcomes such as rehospitalisation, falls, nursing home placement or death has not been sufficiently investigated in the German health and social care system. The few available studies show that interventions related to the home environment can have positive effects on activities of daily living, fall risk and mental health. As the functional abilities of older patients are usually worse at the time of discharge than before hospitalisation, this is a good time to assess the home environment and the person-environment fit.

Integrating professional housing counselling into discharge management could make a significant contribution to increasing safety in the home environment, improving self-help skills and preventing falls and re-hospitalisation. This could improve quality of life and reduce the burden on the healthcare system. The Frail@Home trial is a single-centre, randomised, controlled pragmatic trial (RCT) to test whether housing counselling provided within two to four weeks of hospital discharge increases the chances of older people remaining in their familiar home environment. The intervention group will receive on-site housing counseling, while the control group will receive standard care plus an additional information booklet from the local housing counseling service. The primary endpoint of the study is the number of days spent at home (DSH) in the first 6 and 12 months after discharge from acute geriatric care. The follow-up period will be 12 months. If successful, this study will be the first to show, using RCT methods, that early housing counselling after hospital discharge supports the retention of geriatric patients in their familiar homes.

ELIGIBILITY:
Inclusion criteria:

- Patients aged 70 and over who have been living at home up to now, with typical geriatric multimorbidity and a Barthel Index < 70, who have been admitted to the Wolgast Centre for Geriatric Medicine and whose discharge destination is their own home again. The latter must be in the catchment area of the Wolgast Hospital.

Exclusion criteria:

* Persons who are not able to understand the purpose of the study or who are not able to conduct business (e.g. severe dementia, delirium)
* Patients in a palliative state in the terminal stage
* Patients who are being discharged to a nursing home

T

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Days spent at home 1 year after discharge from geriatrics department | 12 months
  Sum of days spent at home 1 year after discharge from geriatrics department

IPD SHARING:
Plan to Share IPD: Undecided